CLINICAL TRIAL: NCT02606552
Title: Safety and Efficacy of Left Atrial Appendage Closure Versus Antithrombotic Therapy in Patients With Atrial Fibrillation Undergoing Drug-Eluting Stent Implantation Due to Complex Coronary Artery Disease
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The number of patients registered for the study was low and it was expected to be difficult to derive the study results.
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-2014-0074
Record Dates: First submitted 2015-11-12; First posted 2015-11-17 (Estimated); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Atrial Fibrillation; Coronary Artery Disease
Keywords: drug eluting stent; atrial appendage closure
MeSH Terms: conditions — Atrial Fibrillation; Coronary Artery Disease | interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dabigatran plus aspirin (Active Comparator): Medical treatment with dabigatran plus aspirin after 3months triple therapy (Dabigatran plus DAPT (dual-antiplatelet therapy))
  Interventions: Drug: Dabigatrain plus aspirin
- Dabigatran plus clopidogrel (Experimental): medical treatment with dabigatran plus clopidogrel after 3months triple therapy (Dabigatran plus DAPT)
  Interventions: Drug: Dabigatrain plus clopidogrel
- Amplazter Cardiac Plug (ACP) (Other): Amplazter Cardiac Plug (ACP) device-using percutaneous left atrial appendage closure
  Interventions: Device: Amplazter Cardiac Plug (ACP)

INTERVENTIONS:
Drug: Dabigatrain plus aspirin — Dabigatran (Pradaxa®) is indicated for the prevention of thrombotic events (for example stroke or heart attack) in people with atrial fibrillation. Aspirin is indicated for the prevention of stent thrombosis and myocardial infarction in patients treated with drug-eluting stents. Patients will be randomized to stop clopidogrel (maintain dabigatran + aspirin) at 3 months after PCI.
  Arms: Dabigatran plus aspirin
Drug: Dabigatrain plus clopidogrel — Clopidogrel is indicated for the prevention of stent thrombosis and myocardial infarction in patients treated with drug-eluting stents. Patients will be randomized to stop aspirin (maintain dabigatran + clopidogrel) at 3 months after PCI.
  Arms: Dabigatran plus clopidogrel
Device: Amplazter Cardiac Plug (ACP) — Patients allocated to the intervention group should be received percutaneous closure of the LAA by use of the ACP device (St. Jude Medical, St Paul, MN, USA).
  Arms: Amplazter Cardiac Plug (ACP)

SUMMARY:
Comparatively analyze the safety and validity of Amplazter Cardiac Plug (ACP) device-using percutaneous left atrial appendage closure, and the medical treatment with dabigatran plus aspirin or dabigatran plus clopidogrel after 3months triple therapy (Dabigatran plus DAPT (dual-antiplatelet therapy)) in patient with coronary artery disease treated with drug-eluting stent, accompanying atrial fibrillation.

Total of 670 patients [left atrial appendage occlusion registry with 100 ACP/ 570 anti-coagulation registry: (285 Dabigatran plus aspirin) and (285 Dabigatran plus clopidogrel) therapy)] will be comparatively analyzed the safety and efficacy. Primary endpoints were a composite of death, non-fatal myocardial infarction, stroke, systemic embolism, and GUSTO bleeding (moderate to severe).

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 20 years accompanying chronic atrial fibrillation with CHADS2 score ≥2
2. Patients with coronary artery disease (which requires DES) should receive the 2nd generation drug-eluting stent insertion treatment
3. Subjects and their legal representatives must understand the main purpose of this study, agree with relevant provisions, and sign to consent forms approved by IRBs of each institution.
4. Subjects should agree with the follow-up studies as (coronary angiography) and transesophageal echocardiography, etc.
5. Subjects should agree to follow our requests for post-operative follow-up visits.

Exclusion Criteria:

1. Patients showing any hypersensitive reaction or reason for restriction to aspirin, heparin, clopidogrel, or warfarin, or otherwise, susceptible to contrast media, and therefore, who could not use those drugs and who were pregnant or breast feeding.
2. Comorbidities other than atrial fibrillation that required chronic warfarin use.
3. Patients diagnosed with progressive infection condition or endocarditis.
4. Patients who have been diagnosed with progressive gastric ulcer or upper gastrointestinal bleeding for last 3 months.
5. Hemodynamically unstable patients who needs inotropic supports.
6. Senile dementia patients who have experienced any cerebrovascular accident (CVA) for last 6 weeks.
7. Patients who have been diagnosed with intracardiac mass, thrombus, or vegetation as echocardiographic findings.
8. Patients diagnosed with severe left ventricular dysfunction (<LVEF 30%).
9. Patients with blood disorder as followings: leucopenia (<WBC 3,000mm3), acute anemia (<Hg 9mg %), Thrombocytopenia (<100,000 platelets/mm3), or any evidence of bleeding or clotting disorders.
10. Patients showing life expectancy less than 12 months because of noncardiac comorbidities.
11. Patients having severe vein occlusion at femoral vein, ceiling vein, or inferior vena cava.
12. A patent foramen ovale with atrial septal aneurysm and right-to-left shunt
13. Symptomatic carotid artery disease
14. Patients with severe valvular heart disease
15. Patients who are currently participating in other clinical trials for any drug or medical device.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-07-20; Primary Completion 2017-06-23 (Actual); Study Completion 2017-06-23 (Actual)

PRIMARY OUTCOMES:
MACCE (Major adverse cardiac and cerebrovascular events) | 5 years
GUSTO bleeding | 5 years

SECONDARY OUTCOMES:
Occurence of procedural related complications | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Severance Cardiovascular Hospital, Seoul, South Korea